CLINICAL TRIAL: NCT01139489
Title: Stop Antibiotics on Procalcitonin Guidance Study
Brief Title: Safety and Efficacy of Procalcitonin Guided Antibiotic Therapy in Adult Intensive Care Units (ICU's)
Acronym: SAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: UMC Utrecht (Other); Elisabeth-TweeSteden Ziekenhuis (Other); Diakonessenhuis, Utrecht (Other); Isala (Other); Atrium Medical Center (Other); Dijklander Ziekenhuis (Other); Bronovo Hospital (Other); Medical Center Haaglanden (Other); Slotervaart Hospital (Other); University of Groningen (Other); Martini Hospital Groningen (Other); Canisius-Wilhelmina Hospital (Other); Medisch Spectrum Twente (Other); St. Lucas Andreas Ziekenhuis Hospital (Other)
Responsible Party: Principal Investigator, Evelien de Jong, drs, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VU University medical center; NTR1861 (Other: Nederlands Trial Register)
Record Dates: First submitted 2010-03-08; First posted 2010-06-08 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Sepsis; Severe Sepsis; Septic Shock
Keywords: Procalcitonin; antibiotic therapy; antibiotics; sepsis; infections; biomarker
MeSH Terms: conditions — Sepsis; Shock, Septic; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- procalcitonin-guidance (Active Comparator): A daily advise to continue or stop antibiotics based on the measurement of the biomarker procalcitonin
  Interventions: Other: procalcitonin-guidance
- standard-of-care (No Intervention): standard-of-care treatment of ICU infections based upon consensus guidelines and expert opinion

INTERVENTIONS:
Other: procalcitonin-guidance — If procalcitonin levels decrease to predefined levels, antibiotic therapy will be discontinued.
  Other Names: PCT
  Arms: procalcitonin-guidance

SUMMARY:
This is a randomized controlled trial comparing standard-of-care therapy of infections in critically ill patients with a procalcitonin-guided approach evaluating efficacy (antibiotics consumption) and safety (mortality).

DETAILED DESCRIPTION:
Antibiotics are prescribed widely in intensive care units and are linked with high costs and the occurence of antimicrobial (multi)resistance. The optimal duration of antibiotic treatment is poorly known and often based on consensus guidelines.

SAPS is a multicenter, prospective, randomized, controlled open-label trial evaluating the equivalence/efficacy and safety of procalcitonin-guided treatment of infections in ICU patients versus a standard-of-care approach.

All patients that are admitted to the ICU and for whom systemic antibiotics are prescribed for presumed or proven bacterial infections are eligible for this trial. Patients will be randomized and stratified according to clinical diagnosis of severe sepsis and septic shock. Any patient over the age of 18, admitted to the ICU and receiving antibiotics for an assumed infection can be enrolled into this trial. Informed consent has to be obtained in writing from the patient of his/her relatives prior to inclusion. In the intervention group daily procalcitonin levels be performed and will generate a non-binding stopping advice when predefined stopping-rules have been reached. The ultimate decision to stop antibiotics will be at the discretion of the physician in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* receiving antibiotics for no more than 24 hours for an assumed or proven infection
* Informed consent

Exclusion Criteria:

* Failure to obtain written consent to participate
* Patients receiving prolonged antibiotic therapies (> 3 weeks, e.g. endocarditis, cerebral/hepatic abscess)
* Patients with severe infections due to viruses or parasites (e.g. Dengue, Toxoplasma gondii, Plasmodium spp.)
* Patients infected with Mycobacterium tuberculosis
* Patients entering the ICU for post-operative observation and/or on antibiotic prophylaxis with an estimated length of stay less then 24 hrs.
* Patients suffering from cystic fibrosis
* Severely immunocompromised patients such as patients with HIV and with a CD4 count of less than 200 cells/mm, neutropenic patients (<500 neutrophils per mL) or patients with solid organ transplantation
* Moribund patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1575 (Actual)
Dates: Start 2009-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 days
Consumption of antibiotics expressed as the Defined Daily Dosage and duration of antibiotic therapy expressed in days of therapy. | Between day 1 and D28
Mortality | 1 year

SECONDARY OUTCOMES:
Length of ICU stay | Between D1 and D28
Acquisition costs of antibiotics | Between D1-D28
  Expressed in euro's
Acquisition costs of procalcitonin | Between D1-D28
  Expressed in euro's

CONTACTS AND LOCATIONS:
Overall Officials: Evelien de Jong, MSc, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University medical center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Shajiei A, Berends MS, Luz CF, van Oers JA, Harmsen HJM, Vos P, Klont R, Loef BG, Reidinga AC, Bormans-Russell L, Linsen K, Dormans T, Otten M, van der Bij A, Beishuizen A, de Lange DW, de Jong E, Nijsten MW. Impact of reduced antibiotic treatment duration on antimicrobial resistance in critically ill patients in the randomized controlled SAPS-trial. Front Med (Lausanne). 2023 Feb 2;10:1080007. doi: 10.3389/fmed.2023.1080007. eCollection 2023. PMID 36817782
- [Derived] de Jong E, van Oers JA, Beishuizen A, Vos P, Vermeijden WJ, Haas LE, Loef BG, Dormans T, van Melsen GC, Kluiters YC, Kemperman H, van den Elsen MJ, Schouten JA, Streefkerk JO, Krabbe HG, Kieft H, Kluge GH, van Dam VC, van Pelt J, Bormans L, Otten MB, Reidinga AC, Endeman H, Twisk JW, van de Garde EMW, de Smet AMGA, Kesecioglu J, Girbes AR, Nijsten MW, de Lange DW. Efficacy and safety of procalcitonin guidance in reducing the duration of antibiotic treatment in critically ill patients: a randomised, controlled, open-label trial. Lancet Infect Dis. 2016 Jul;16(7):819-827. doi: 10.1016/S1473-3099(16)00053-0. Epub 2016 Mar 2. PMID 26947523
- [Derived] Assink-de Jong E, de Lange DW, van Oers JA, Nijsten MW, Twisk JW, Beishuizen A. Stop Antibiotics on guidance of Procalcitonin Study (SAPS): a randomised prospective multicenter investigator-initiated trial to analyse whether daily measurements of procalcitonin versus a standard-of-care approach can safely shorten antibiotic duration in intensive care unit patients--calculated sample size: 1816 patients. BMC Infect Dis. 2013 Apr 16;13:178. doi: 10.1186/1471-2334-13-178. PMID 23590389